CLINICAL TRIAL: NCT05837481
Title: Decreasing Sedative Requirements for Peripheral Vascular Interventions Using Preoperative Guided Meditation
Brief Title: Guided Meditation to Decrease Perioperative Anxiety and Increase Patient Intraoperative Compliance in Vascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anahita Dua, MBCHB, MBA, MSC, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P002072; F32HS028943-01 (AHRQ)
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Meditation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The proceduralists that will be performing the peripheral vascular interventions will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group (Experimental): Two sessions of guided meditation on the day of surgery, both to occur before the start of surgery
  Interventions: Behavioral: Meditation
- Control Group (No Intervention): Standard of care, which does not involve any meditation programs

INTERVENTIONS:
Behavioral: Meditation — Guided meditation utilizing breath awareness, body scan and visualization techniques
  Arms: Meditation Group

SUMMARY:
The primary purpose of this clinical trial is to test the feasibility of implementing a perioperative guided meditation program for patients undergoing peripheral vascular interventions that are performed under procedural sedation and analgesia.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled study involving 30 adult patients undergoing peripheral vascular interventions. Patients will be randomized to two arms: an intervention arm where patients will participate in perioperative guided meditation, and a control arm where patients will receive standard of care without any meditation intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing an endovascular procedure for peripheral vascular disease
* Anesthesia plan for procedural sedation and analgesia

Exclusion Criteria:

* Pre-existing psychiatric disorder such as anxiety, panic disorder, depression, psychosis, or bipolar disorder
* Non-English speaking
* Prior history of ipsilateral lower extremity amputation
* Urgent or Emergent Surgery
* Anesthesia plan for general anesthesia
* Undergoing a hybrid procedure (simultaneous endovascular and open surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chien Yi M Png, MD, Study Chair — Massachusetts General Hospital; Chien Yi M Png, MD, Study Director — Massachusetts General Hospital; Anahita Dua, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Salem Hospital, Salem, Massachusetts
  - Southern New Hampshire Hospital, Nashua, New Hampshire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meditation Group | Control Group
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — index procedure changed to an open surgical procedure that required general anesthesia. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meditation Group | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (14.9) | 72.3 (9.05) | 71.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
PROMIS-10 Score [Mean (Standard Deviation); unit: score] — The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health survey is a patient-reported measure of health-related quality of life. The score range for the PROMIS-10 is from 0 to 20. Higher scores indicate higher quality of life, and thus are better.
  score | 9.4 (2.35) | 10.2 (2.42) | 9.8 (2.38)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Implementing Preoperative Guided Meditation
Description: Feasibility will be defined as >80% of the patients enrolled in the intervention arm having successfully completed both rounds of perioperative meditation.
Time Frame: Immediately before surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Meditation Group | Control Group
Number analyzed (Participants) | 15 | 14
Participants | 15 | 14

2. Secondary Outcome: Anxiety - STAI-6
Description: The State-Trait Anxiety Inventory (STAI) is a patient-reported measure of anxiety. The score range for the STAI-6 is from 6 to 24. Higher scores indicate higher anxiety, and thus are worse.
Time Frame: Preoperative (prior to meditation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditation Group | Control Group
Number analyzed (Participants) | 15 | 15
units on a scale | 11.93 (4.43) | 11.86 (3.94)

3. Secondary Outcome: Interoceptive Attention - MAIA (Noticing Sub Scale)
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a patient-reported measure of interoceptive attention. Higher scores indicate higher interoception, and thus are better. This sub scale score represented the combined scores of the 4 questions in the noticing sub scale, and ranged from 0 to 20.
Time Frame: Preoperative (prior to meditation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditation Group | Control Group
Number analyzed (Participants) | 15 | 15
units on a scale | 12.8 (5.08) | 10.7 (4.87)

4. Secondary Outcome: Anxiety - STAI-6
Description: as for outcome 2
Time Frame: Postoperative (within 6 hours after surgery)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditation Group | Control Group
Number analyzed (Participants) | 15 | 14
units on a scale | 8.33 (2.22) | 9.42 (3.39)

5. Secondary Outcome: Interoceptive Attention - MAIA (Noticing Sub Scale)
Description: as for outcome 3
Time Frame: Postoperative (within 6 hours after surgery)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditation Group | Control Group
Number analyzed (Participants) | 15 | 14
units on a scale | 14.3 (4.46) | 11.5 (4.92)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment until the completion of the perioperative meditation program.
Arm/Group | Meditation Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT05837481/Prot_SAP_000.pdf